CLINICAL TRIAL: NCT05477355
Title: Increasing Mental Health and Psychosocial Social Support for Venezuelan Refugees and Migrants: Adapting Group Problem Management Plus (Group PM+) for Venezuelan Refugees and Migrants in Colombia
Brief Title: Adapting Group PM+ for Venezuelan Refugees and Migrants in Colombia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The New School (Other)
Collaborators: Universidad del Norte (Other); Columbia University (Other); HIAS (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: GR20920
Record Dates: First submitted 2022-07-19; First posted 2022-07-28 (Actual); Last update posted 2022-07-28 (Actual); Status verified 2022-07

CONDITIONS: Mental Health Wellness 1

STUDY DESIGN:
Intervention Model Description: The intervention is Group Problem Management Plus (PM+).
Masking Description: Participants in wait list control (WLC) are explained that they will be receiving the intervention at a later time.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Experimental): Participants will be provided the 5 session intervention.
  Interventions: Behavioral: Group Problem Management Plus (PM+)
- Wait list control arm (Active Comparator): Participants will not be provided Group PM+ in Phase 1 but will be provided the intervention after all participants in the initial intervention arm receive Group PM+.
  Interventions: Behavioral: Group Problem Management Plus (PM+)

INTERVENTIONS:
Behavioral: Group Problem Management Plus (PM+) — Group PM+ is a low-intensity, trans-diagnostic, brief psychological intervention developed by the WHO. Group PM+ consists of five sessions delivered in five consecutive weeks and includes strategies that are aimed towards decreasing symptoms of depression, anxiety, general distress, and other related conditions. Group PM+ is designed to be delivered by non-specialists, persons without a formal education and licensure in psychology or mental health.

SUMMARY:
This study is a type 2 hybrid implementation design, which aims to evaluate the utility and effectiveness of an intervention while simultaneously assessing implementation outcomes, such as adoption, fidelity, and maintenance. The aim is to compare participant level outcomes when the intervention is delivered by facilitators that are trained and supervised by psychologists versus by lay-supervisors. Group PM+ will be delivered to participants in two phases: first, with high levels of technical support through intensive training and supervision by mental health professionals and a second phase with routine service delivery and supervision. Non-specialist community members who are trained and supervised by psychologists to deliver PM+ as part of Phase 1 will be trained to become supervisors and train and support a cohort of new non-specialist facilitators for Group PM+ delivery in Phase 2. This model employs a train-the-trainers model to replicate routine service delivery especially in settings where mental health specialists may not be available to provide robust technical support and supervision to lay PM+ facilitators. The aim is to compare effectiveness and implementation outcomes of Group PM+ when delivered within routine care, to identify best practices for implementation, and ultimately, to shorten the time lag between intervention research and routine uptake.

DETAILED DESCRIPTION:
This study is a type 2 hybrid implementation design, which aims to evaluate the utility and effectiveness of an intervention while simultaneously assessing implementation outcomes, such as adoption, fidelity, and maintenance. The aim is to compare participant level outcomes when the intervention is delivered by facilitators that are trained and supervised by psychologists versus by lay-supervisors. Group PM+ will be delivered to participants in two phases: first, with high levels of technical support through intensive training and supervision by mental health professionals and a second phase with routine service delivery and supervision. Non-specialist community members who are trained and supervised by psychologists to deliver PM+ as part of Phase 1 will be trained to become supervisors and train and support a cohort of new non-specialist facilitators for Group PM+ delivery in Phase 2. This model employs a train-the-trainers model to replicate routine service delivery especially in settings where mental health specialists may not be available to provide robust technical support and supervision to lay PM+ facilitators. The aim is to compare effectiveness and implementation outcomes of Group PM+ when delivered within routine care, to identify best practices for implementation, and ultimately, to shorten the time lag between intervention research and routine uptake.

This research design offers a few points of comparison:

1. change in primary and secondary outcomes at 1-week follow-up and 3-month follow-up amongst participants that receive Group PM+ with research support (Phase 1) compared to those that receive the intervention with standard care and implementation (Phase 2), [Primary objective]
2. differences in implementation indicators (ex. Facilitator competencies, fidelity to PM+, participant retention, cost effectiveness, adverse events, human resource involvement and more) in Phase 1 of implementation compared to Phase 2,
3. change in primary and secondary outcomes amongst participants in the intervention arm compared to participants who do not receive the intervention during Phase 1.

ELIGIBILITY:
Inclusion Criteria:

* must identify as a woman
* over 18 years of age
* must state that they are planning to live in Barranquilla for at least three months after the date of screening
* moderate functional impairment as indicated by scoring greater than 16 on the WHO Disability Assessment Schedule 2.0 (WHODAS 2.0) for health and disability
* moderate psychological distress as indicated by scoring greater than 2 on the General Health Questionnaire 12 (GHQ-12)

Exclusion Criteria:

* imminent risk of suicide and state that they have plans for attempting suicide
* show severe cognitive impairment (e.g. severe intellectual disability or dementia) or a severe disability as identified by the Ten Questions (TQ-10)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Participants that self-identify as women are eligible for the study
Enrollment: 140 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Patient Health Questionnaire 9 (PHQ-9) | 4 months after baseline
  a well-known 10-item instrument that measures symptoms of depression and general distress. It has been used in prior PM+ studies as the primary participant level outcome.
  Scoring between 5-9 points indicates mild depression, 10-14 points indicates moderate depression, 15-19 points indicates moderately severe depression, and 20 or more points indicates severe depression.

SECONDARY OUTCOMES:
Post-traumatic stress disorder Checklist (PCL-5) | 4 months after baseline
  a 20-item checklist that corresponds with the 20 DSM IV PTSD symptoms
Psychological Outcome Profiles (PSCYHLOPS) | 4 months after baseline
  This instrument seeks participants perspectives on their psychological distress related to the problems they are facing and well-being scored on a 0 to 5 scale
Reducing Tension Checklist (RTC) | 4 months after baseline
  12-item assessment of psychological and behavioral skills related to PM+ to evaluate skill acquisition
Alcohol use disorders identification test (AUDIT) | 4 months after baseline
  This assessment measures hazardous and harmful alcohol use.

CONTACTS AND LOCATIONS:
Overall Officials: Adam Brown, PhD, Principal Investigator — The New School
Locations (1):
- HIAS, Barranquilla, Colombia

IPD SHARING:
Plan to Share IPD: No
All participant data will anonymized when input into databases. Individual participant data will only be available to those on the research team.